CLINICAL TRIAL: NCT01655342
Title: Assessment of the Effectiveness of Biodentine® in Pulpotomies Primary Teeth.
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: Moran- HMO-CTIL
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Effectiveness of Biodentine® in Pulpotomies Primary Teeth
Keywords: pulpotomy; primary teeth; Biodentine®; formocresol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- formocresol

SUMMARY:
Clinical and radiographic assessment of Biodentine® as a pulp dressing material for pulpotomy treatment in human primary molars.

ELIGIBILITY:
Inclusion Criteria:

* one or more primary teeth which requires pulpotomy.

Exclusion Criteria:

* not healthy patients,
* patients with teeth which requires pulpectomy.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children attending the Pediatric Dentistry Clinic of the Hebrew University-Hadassah School of Dental Medicine in Jerusalem
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2012-08; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Success of the primary molar pulpotomy | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Laurent P, Camps J, About I. Biodentine(TM) induces TGF-beta1 release from human pulp cells and early dental pulp mineralization. Int Endod J. 2012 May;45(5):439-48. doi: 10.1111/j.1365-2591.2011.01995.x. Epub 2011 Dec 22. PMID 22188368